CLINICAL TRIAL: NCT04158999
Title: Descriptive, Observational, Investigation of the Effect of Mother's Nutrition Status on Breast Milk Contents
Brief Title: Investigation of the Effect of Mother's Nutrition Status on Breast Milk Contents
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Halic University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Fatma Şule Bilgiç, Research Asst., Halic University
Other Study IDs: SuleTez
Record Dates: First submitted 2019-11-04; First posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Breast Feeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Mother milk: Step 1: Mothers who meet the sample selection criteria will be informed about the scope of the study and their written and verbal consent will be obtained. Data collection form will be applied to mothers who accept to participate in the study by using face to face interview technique. Mothers and newborns will be weighed and 4 ml breast milk sample will be taken from the mother for manual milking.
  Interventions: Device: milk analyzer; Behavioral: Mother's nutrition values

INTERVENTIONS:
Device: milk analyzer — Human Milk Sample
  Other Names: Human Milk Sample
Behavioral: Mother's nutrition values — evaluation of nutritional elements of maternal onset with Bebis Program

SUMMARY:
This study; this work; The aim is to investigate the effects of mothers' nutritional status on breast milk macro nutrients (carbohydrate, fat and protein).

DETAILED DESCRIPTION:
Macronutrients in breast milk can be affected by various factors. The mothers will be taken in the first 24 hours after birth and their nutritional habits, socio-demographic characteristics, anthropometric characteristics of the mother, body mass index will be examined and newborn characteristics will be taken. 2 ml sample from colostrum will be analyzed with milk analyzer instrument. The mothers will be re-checked on the 5th day and their anthropometric properties will be obtained. The same procedure will be repeated on the 15th day after childbirth. At each control, the mother's last 24-hour feeding status will be taken and the nutritional values consumed by "BeBis" program will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Follow-up of the infant in the Neonatal Intensive Care Unit, Istanbul Faculty of Medicine, Department of Pediatrics,

  * The mother is able to understand and answer the questions,
  * Single pregnancy,
  * The baby's birth week is 34 weeks or more,
  * The mother does not have a disease (Diabetes, hypertension, hypothyroidism, etc.) that may affect breast milk content.

Exclusion Criteria:

* Multiple pregnancy,

  * The birth week of the baby is less than 34 weeks.
  * Breastfeeding or breast problems in the mother,
  * The mother has a disease that may affect breast milk content (Diabetes, hypertension, hypothyroidism, etc.),
  * The mother is not willing to participate in the research,
  * A disease known to be transmitted by breast milk (HIV, hepatitis B, hepatitis C, etc.).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Mother,postpartum
Study Population: Mothers whose babies were followed in the neonatal follow-up outpatient clinic of the Neonatal Intensive Care Unit of Istanbul University Faculty of Medicine, Department of Pediatrics and Fifty will be composed of 50 mothers who meet the sample selection criteria.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-11-10 (Estimated); Primary Completion 2020-02-12 (Estimated); Study Completion 2020-05-12 (Estimated)

PRIMARY OUTCOMES:
Human Milk Macro Nutrients | 15 Days
  CHA,Protein, Fat

SECONDARY OUTCOMES:
Mother's Diet | 24 hours
  BMI

CONTACTS AND LOCATIONS:
Overall Officials: Gulçin Bozkurt, Assc. Prof., Study Director — Istanvbul University-Cerrahpasa; Asuman Çoban, Prof, Study Director — Istanbul University

IPD SHARING:
Plan to Share IPD: Yes
The population of the study will be composed of mothers whose babies are followed in the neonatal follow-up outpatient clinic of the Neonatal Intensive Care Unit of Istanbul University Faculty of Medicine, Department of Child Health and Diseases.
  data collection form total of 69 questions; women's socio-demographic characteristics11 questions, baby's characteristics and nutrition10 questions, obstetric characteristics of pregnancy, curettage, abortion, childbirth 11 obstetric questions, features related to breastfeeding 8 questions, the mother's feeding habits 5 questions and 24 questions about the results of the mother's milk sample It is a daily (last 24 hours) form of food consumption which is required to indicate the foods consumed in the last 24 hours before. Data collection tools will be applied using face to face interview technique.
Supporting Information: Study Protocol, SAP
Time Frame: 8 mounts
Access Criteria: One year

REFERENCES:
- [Background] Butts CA, Hedderley DI, Herath TD, Paturi G, Glyn-Jones S, Wiens F, Stahl B, Gopal P. Human Milk Composition and Dietary Intakes of Breastfeeding Women of Different Ethnicity from the Manawatu-Wanganui Region of New Zealand. Nutrients. 2018 Sep 4;10(9):1231. doi: 10.3390/nu10091231. PMID 30181524
- [Result] Bravi F, Wiens F, Decarli A, Dal Pont A, Agostoni C, Ferraroni M. Impact of maternal nutrition on breast-milk composition: a systematic review. Am J Clin Nutr. 2016 Sep;104(3):646-62. doi: 10.3945/ajcn.115.120881. Epub 2016 Aug 17. PMID 27534637